CLINICAL TRIAL: NCT05817682
Title: Interprofessional Education of Medical Students Using Medical Simulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Barbara Siekierska, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WLNZ/NoZ/2022
Record Dates: First submitted 2023-03-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Medical Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Interprofessional education
- Control group (No Intervention)

INTERVENTIONS:
Other: Interprofessional education — The study will be conducted among students of the Krakow Academy. The experimental group will consist of 35 students participating in the Interdisciplinary Circle of Medical Simulation from the following faculties: medicine, nursing and medical rescue.
  Students will be divided into 7 interprofessional teams, in which they will take classes planned for small groups.
  Arms: Intervention group

SUMMARY:
Due to the growing role of medical simulation in the education of medical students and the development of cooperation in interdisciplinary teams in the health care sector, a study was designed to examine the relationship between the competences and resources of students and the role of education through simulation classes based on the development of technical and in cooperation with specialists in these fields. Researchers want to focus on students' levels of stress and anxiety, coping strategies, and self-efficacy. An important element will be the self-assessment of students on the level of their non-technical competences.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent to participate in the study
* Declaration of participation in the Interdisciplinary Simulation Circle
* Student status in the field of medicine (6th year) or nursing (3rd year of first-cycle studies) or medical rescue (3rd year)

Exclusion Criteria:

* Completed another course of medical studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the ongoing interprofessional education | 10 months
  1. A self - report questionnaire including a socio-demographic data sheet and questions regarding the motivation for choosing the field of study, as well as a form for the ongoing evaluation of Interdisciplinary Club classes to be completed before and after classes.
Evaluation of the impact of interprofessional education on soft-skill development | 10 months
  1. Self-assessment form in the field of soft skills - own study, which contains 17 statements describing soft skills in an interprofessional team. Respondents assess their development on a five-point Likert scale, where "1" means "I completely disagree" and "5" - "I completely agree".
Evaluation of the impact of interprofessional education using the simulation method on self-efficacy. | 10 months
  1. General Self-Efficacy Scale (GSE) with the total score calculated by finding the sum of all the items and ranges between 10 and 40, with higher score indicating more self-efficacy.
Evaluation of the impact of interprofessional education using the simulation method on student stress level. | 10 month
  A 10-item Perceived Stress Scale (PSS-10) for assessing how often a respondent thought and felt in the given way in the last month using a five-point Likert scale. The result of the measurement is the stress severity index. The PSS score is obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
Evaluation of the impact of interprofessional education using the simulation method on stress coping. | 10 month
  The Stress Coping Inventory (Mini COPE). The respondent determines how often he/she acts in the described way when experiencing a stressful situation using a four-point Likert scale (0-I almost never do that, 1-I rarely do that, 2-I often do that, 3-I almost always do that). Every statement is assigned to one of 14 stress-coping categories.
Evaluation of the impact of interprofessional education using the simulation method on perception of medical professions. | 10 month
  Word Cloud - own study - a form used to assess the mutual perception of medical professions in an interprofessional team. The respondents choose five terms from the proposed word database.
Evaluation of the impact of interprofessional education using the simulation method on students anxiety. | 10 month
  A 20-item State-Trait Anxiety Inventory (STAI) for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrzej Frycz Modrzewski Krakow University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided